CLINICAL TRIAL: NCT01522196
Title: A Randomized, Double-blind, Placebo-Controlled Study With Varespladib Infusion (A-001) in Subjects With Sickle Cell Disease and Vaso-Occlusive Crisis for the Prevention of Acute Chest Syndrome At-Risk Subjects.
Brief Title: A Study of Varespladib Infusion in Subjects With Sickle Cell Disease.
Acronym: IMPACTS-2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: change in company plans
Sponsor: Anthera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AN-SCD1122
Record Dates: First submitted 2012-01-18; First posted 2012-01-31 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-01

CONDITIONS: Sickle Cell Disease; Vaso-occlusive Crisis
Keywords: SCD
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises | interventions — varespladib; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Varespladib (Active Comparator): 48 hour continuous infusion delivered intravenously (IV)
  Interventions: Drug: Varespladib
- Placebo (Placebo Comparator): 48 hour continuous infusion delivered intravenously (IV)
  Interventions: Other: Placebo (Normal Saline)

INTERVENTIONS:
Drug: Varespladib — 48 hour continuous infusion delivered intravenously (IV)at a rate of 110µg/kg/hr.
  Arms: Varespladib
Other: Placebo (Normal Saline) — 48 hour continuous infusion delivered intravenously (IV)at a rate of 110µg/kg/hr.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effectiveness of A 001 infusion in preventing acute chest syndrome in sickle cell disease (SCD) subjects with vaso-occlusive crisis, fever, and elevated serum C-reactive protein (CRP).

ELIGIBILITY:
Inclusion Criteria:

* Genotypes Hb SS, Hb SC, sickle β°-thalassemia, sickle β+ -thalassemia
* Pain consistent with vaso-occlusive crisis (clinical judgment) and not attributable to other causes
* Serum CRP ≥5.0 mg/L at time of screening
* Fever defined as oral temperature ≥38.0°C at time of screening
* Age ≥5 years

Exclusion Criteria:

* New or suspected new pulmonary infiltrate diagnosed by chest radiography
* Females who are nursing, pregnant or intend to become pregnant
* Renal dysfunction defined as a creatinine level >1.2 mg/dL for subjects aged 18 or less or a creatinine level >1.5 mg/dL for subjects over the age of 18
* Hepatic dysfunction (alanine aminotransferase [ALT] or aspartate aminotransferase [AST] >3 × upper limit of normal)
* Acute neurologic dysfunction
* Any medical condition for which transfusion may be needed imminently, and/or hemoglobin <5 g/dL
* Red blood cell transfusion within 30 days prior to screening
* Parenteral or oral corticosteroid therapy (inhaled steroids acceptable) within 7 days prior to screening

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Efficacy of A 001 infusion in preventing acute chest syndrome in sickle cell disease (SCD) subjects with the combination of vaso-occlusive crisis, fever, and elevated serum C-reactive protein (CRP). | Various time points up to Day 30

SECONDARY OUTCOMES:
Safety and tolerability of A 001 therapy when administered as a 48-hour continuous infusion to SCD subjects at-risk for acute chest syndrome. | Various time points up to Day 30
Impact of A-001 treatment on sPLA2 levels and CRP. | Various time points up to Day 30
Impact of A-001 treatment on the signs and symptoms of vaso-occlusive crisis. | Various time points up to Day 30
Impact of A-001 treatment on opioid use for pain in the treatment of vaso-occlusive crisis. | Various time points up to Day 30

CONTACTS AND LOCATIONS:
Locations (1):
- Investigator Site 101, Atlanta, Georgia, United States